CLINICAL TRIAL: NCT04500847
Title: Repurposing Nucleoside Reverse Transcriptase Inhibitors for Treatment of AD
Acronym: LINE-AD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Alzheimer's Association (Other); Brown University (Other); The Miriam Hospital (Other); Cedars Sinai Medical Center, Los Angeles, USA (Unknown)
Responsible Party: Principal Investigator, Meghan Riddle, Director of Neurology and the Memory and Aging Program, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LINE-AD
Record Dates: First submitted 2020-06-15; First posted 2020-08-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease, Early Onset; Mild Cognitive Impairment; Moderate Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Emtricitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist will not be masked. All investigators will be masked until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): 25 MCI and mild to moderate AD subjects
  Interventions: Drug: Emtriva Capsule
- Group 2 (Placebo Comparator): 10 MCI and mild to moderate AD subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emtriva Capsule — 200mg daily oral dose
  Other Names: Emtricitabine
  Arms: Group 1
Drug: Placebo — 200mg daily oral dose
  Other Names: Capsule manufactured to mimic Emtriva
  Arms: Group 2

SUMMARY:
This is a randomized, double-blind clinical trial of a daily oral dose of 200 mg emtricitabine vs. placebo in 35 participants with biomarker-confirmed MCI or mild to moderate dementia due to Alzheimer's disease. Study duration for each subject participating in the placebo-controlled research study will be approximately 12 months (up to a 3 months Screening Period, Baseline visit (1 month), 6 months of placebo or emtricitabine dosing, and 1 month follow-up). Participants will have up to 2 months to complete all procedures for the month 6 study visit.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a devastating and increasingly frequent neurological disorder whose onset is strongly correlated with advanced age. Between 2000 and 2017 deaths from AD have increased 145%, and AD has become the 6th leading cause of death in the USA. Unfortunately, in spite of immense research and clinical efforts spanning several decades, cures have been elusive. This has prompted searches for new mechanisms of disease and new targets of therapy. One such direction is inflammation: aging and many age-associated diseases are believed to be causally linked with a chronic inflammatory state. The brain is no exception, and the presence of inflammation in the AD brain establishes an environment that is hostile for the function and survival of neurons. While it is not yet clear whether inflammation is the root cause of AD, it is increasingly believed that alleviating these inflammatory processes might slow down the progression of the disease. This research study will test to determine if the inflammatory state can be alleviated with a class of drugs known as nucleoside reverse transcriptase inhibitors (NRTIs). NRTIs were developed to treat Acquired Immune Deficiency Syndrome (AIDS) caused by infection with Human Immunodeficiency Virus (HIV). Investigators hypothesize that NRTI drugs, by inhibiting neuroinflammation, may be effective in the treatment of AD. The primary goal of this trial will be to assess safety and tolerability of Emtriva in a geriatric population of individuals diagnosed with mild cognitive impairment or early AD.

This study will be conducted in subjects with mild to moderate Alzheimer's disease (AD), including subjects with mild cognitive impairment (MCI). Subjects must be positive for amyloid pathology. Subjects must be 50 to 85 years old, and apart from the clinical diagnosis of early AD, in good health as determined by the Investigator based on their medical history. Participants must be HIV/HBV negative and pass all the screening assessments based on the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 50-85 years inclusive
* Intellectually, visually and auditory capable, fluent in, and able to read, the language in which study assessments are administered (e.g. completion of at least six years of regular schooling or sustained employment or equivalent local level of knowledge).
* Must meet NIA-AA research criteria for MCI and mild dementia due to AD
* Mini Mental State Exam (MMSE) 15-30 inclusive
* Clinical Dementia Rating (CDR) 0.5 - 2
* Must meet a cerebrospinal fluid (CSF) pTau/Aβ42 ratio of > 0.024
* Participants must have an appropriate study partner who agrees to participate in the study and who is intellectually, visually, and auditory capable, and fluent in, and able to read, the language in which study assessments are administered. Additionally, the study partner must be capable of and willing to: Accompany the participant to visits that requires the input of the study partner
* Concurrent treatment with cholinesterase inhibitors and memantine are permitted on a stable dose for at least 60 days prior to baseline.

Exclusion Criteria:

* Current medical or neurological condition that might impact cognition or performance on cognitive assessments, e.g., Huntington's disease, Parkinson's disease, syphilis, schizophrenia, bipolar disorder, active major depression, attention deficit/ hyperactivity disorder (ADD/ADHD), multiple sclerosis (MS), amyotrophic lateral sclerosis (ALS), active seizure disorder, current alcohol/drug abuse or dependence, or dependence within the last two years, or history of traumatic brain injury associated with loss of consciousness and ongoing residual transient or permanent neurological signs/symptoms including cognitive deficits, and/or associated with skull fracture
* Brain MRI results showing findings unrelated to AD that, in the opinion of the investigator might be a leading cause of future cognitive decline, might pose a risk to the participant, or might confound MRI assessment for safety monitoring
* Score "yes" on item four or item five of the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale (eC-SSRS patient-reported outcome), if this ideation occurred in the past six months, or "yes" on any item of the Suicidal Behavior section, except for the "Non-Suicidal Self-Injurious Behavior" (item is included in the Suicidal Behavior section), if this behavior occurred in the past 2 years prior to screening
* Use of other investigational drugs prior to screening until:

  * Small molecules: after five half-lives, or within 30 days until the expected pharmacodynamic effect has returned to baseline, whichever is longer
  * Biologicals: blood concentration has returned to baseline (or below serological responder threshold) for antibodies induced by active immunotherapy; or five half- lives for monoclonal antibodies or other biologicals
* Approximately four weeks prior to randomization, the use of any drug or treatment known for the potential to cause major organ system toxicity, i.e. drugs that may require periodic safety monitoring of a specific organ or body fluid. Examples include, but are not limited to clozapine, cancer medical treatment like tamoxifen, systemic immunosuppressive drugs like methotrexate or interferon, or other immunosuppressive biological medicines for rheumatic diseases or multiple sclerosis
* A positive drug screen, if, in the investigator's opinion, this is due to drug abuse or dependence.
* Significant ECG findings that are assessed as clinically significant by the investigator (e.g. sustained ventricular tachycardia, significant second or third degree atrioventricular block without a pacemaker, long QT syndrome or clinically meaningful prolonged QT interval).
* Contraindication to lumbar puncture including use of anti-coagulants, low platelet count, history of back surgery (with the exception of microdiscectomy or laminectomy over one level), signs or symptoms of intracranial pressure, spinal deformities or other spinal conditions that in the judgment of the investigator would preclude a lumbar puncture
* History of or active hepatitis or HIV infection (based on a positive lab result for HBV and/or HIV, to be performed during screening
* Severe renal impairment
* Severe hepatic impairment
* Significant cardiac disease including recent (within six months) myocardial infarction, congestive heart failure or unstable angina
* Female subjects who are pregnant or currently breastfeeding.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAE's) in the treatment group will be compared to the placebo group | Baseline to the follow up study visit (7-8 months after first treatment)
  Number of participants with treatment emergent adverse events and serious adverse events as assessed by CTCAE (Version 4.03).

SECONDARY OUTCOMES:
Change from baseline in key inflammatory biomarkers; Tumor necrosis factor-alpha (TNF-α), Interleukin 1-beta (IL-1β), and Interferon-alpha (IFN-α) | Baseline to the follow up study visit (7-8 months after first treatment)
  Blood draws will be taken from baseline to the follow up study visit. Inflammation and discovery research assays to detect levels of TNF-α, IL-1β, and IFN-α will be performed at Brown University.
Change in Mini Mental State Examination (MMSE) Total Scores | Screening phase, month 3 and month 6 after first treatment
  To determine changes of the MMSE scores from the screening phase to 6 months after first treatment.
Change from baseline in Clinical Dementia Rating (CDR) | Screening phase, month 3 and 6 months after first treatment
  To determine changes of CDR scores from screening phase to 6 months after first treatment.
Change from baseline in Alzheimer's Disease Assessment Scale-cognitive (ADAS-Cog -13) | Screening phase, month 3 and month 6 after first treatment
  To determine changes in ADAS-Cog scores from screening phase to 6 months after first treatment.
Change from baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | Screening phase, month 3 and month 6 after first treatment
  To determine changes in ADCS-ADL scores from screening phase to 6 months after first treatment.
Change from baseline in Free and Cued Selective Reminding Test (FCSRT+IR) with delayed recall | Screening phase, month 3 and month 6 after first treatment
  To determine changes in FCSRT+IR with delayed recall from screening phase to 6 months after first treatment.
Change from baseline in cerebrospinal fluid (CSF) phosphorylated tau/amyloid beta 42 (pTau/Aβ42) ratios | Screening phase to month 6-7 after first treatment
  To determine changes in pTau/Aβ42 ratios from the screening phase to 6 months after first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Riddle, MD, Principal Investigator — Butler Hospital; John Sedivy, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Memory and Aging Program, Butler Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez P, Zuniga G, Sun W, Beckmann A, Ochoa E, DeVos SL, Hyman B, Chiu G, Roy ER, Cao W, Orr M, Buggia-Prevot V, Ray WJ, Frost B. Pathogenic tau accelerates aging-associated activation of transposable elements in the mouse central nervous system. Prog Neurobiol. 2022 Jan;208:102181. doi: 10.1016/j.pneurobio.2021.102181. Epub 2021 Oct 17. PMID 34670118